CLINICAL TRIAL: NCT01939769
Title: Acute Effects of Exercise on Memory in Healthy and Brain-Injured Individuals
Brief Title: Effects of Exercise on Memory in Healthy and Brain-Injured Individuals
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 130198; 13-N-0198
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08-28

CONDITIONS: Traumatic Brain Injury
Keywords: fMRI; Catecholamines; Stress; Exercise; Memory
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity | interventions — High-Intensity Interval Training

INTERVENTIONS:
Other: Exercise - Low-intensity exercise
Other: Exercise - High-intensity exercise

SUMMARY:
Background:

- Research has shown that one exercise session may improve a person s ability to recall information they learned before the exercise. Knowing how exercise changes brain activity to improve memory can help researchers understand how memory works and how to improve it in people with memory problems. This study compares two kinds of exercise on a stationary bike for their ability to temporarily improve memory on certain tests. Researchers will look at the effect of exercise on body chemistry by drawing blood and collecting saliva.

Objectives:

- To understand how a single session of exercise affects memory testing in healthy people and people who have had traumatic brain injury (TBI).

Eligibility:

* Adults ages 18 through 45 with TBI.
* Healthy adult volunteers, ages 18 through 45.

Design:

* Participants will be screened with medical history and physical exam. This will take about 1 hour.
* Participants with TBI will also be screened with a test of their memory. This will take another hour.
* Visit 1 will take about 3 hours. Participants will:

<TAB>- Have a tube inserted in their arm for drawing blood during the tests.

<TAB>- Take memory tests. They will look at pictures, symbols, and words, then answer questions.

<TAB>- Give a saliva sample by chewing on a small sponge for 2 minutes.

<TAB>- Exercise on a stationary bike.

<TAB>- Take the memory tests again.

- Visit 2 will take place 1 week later. Participants will take the memory tests only.

DETAILED DESCRIPTION:
Objective: The goals of this study are to 1. replicate the finding that exercise after exposure to images enhances their subsequent recall, 2. extend the question to words and logical rules, 3. examine the mechanism of the effect using exercise biomarkers and fMRI and 4. explore its usefulness as an aid to memory in individuals with traumatic brain injury (TBI).

Study population: Healthy adult volunteers and individuals with TBI.

Design: The main, clinical, experiment has a parallel, repeated-measures design, where four groups (two each of healthy subjects and participants with TBI) will encode pictures, words and rules and then exercise at either a high or very low (placebo) intensity. Recall will be tested one hour and again at seven days after exercise. Blood and saliva will be collected before and immediately after exercise and assayed for biomarkers of exercise, thought to be possible mediators of the memory effect. In a parallel-design fMRI experiment, intended to explore the brain basis of the effect of exercise on memory, healthy volunteers will view pictures, exercise at a high or low intensity, and then perform a recall task in the scanner. The analysis will look for differences in location and extent of evoked brain activations evoked by picture recall after low and high intensity exercise.

Outcome measures: The primary outcome measure is recall of visual material one hour after exercise. Secondary measures will be the recall of word lists and letter/digit symbol matching (logical memory) and activations on fMRI. The blood and saliva biomarkers will are included as exploratory outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:

<TAB>

* Age 18-45 (inclusive)
* English speaking and writing
* For TBI patients:<TAB>

  * History of TBI (defined according to the American Congress of Rehabilitation Medicine Criteria: History of having sustained a traumatically induced physiological disruption of brain function at least 2 months before participation)
  * Evidence of at least moderate TBI severity. Evidence for intensity of TBI will be any one of the following 3 criteria:

    1. GCS greater than or equal to 9 (obtained in Emergency Room and noted in medical record)
    2. Post-traumatic amnesia > 24 hours
    3. TBI-related abnormality on neuroimaging (either CT or MRI)
  * Documented memory deficit, i.e., a score of 1 standard deviation or more below age-adjusted norm on a recognized clinical test of memory, such as the Wexler Memory Scale, within the last two years.
  * Enrollment in Protocol 11-N-0084
* Right-handedness for fMRI participants

EXCLUSION CRITERIA:

* Inability to give informed consent
* History of major neurological or psychiatric illness, e.g., neurodegenerative disorder, stroke, congenital or genetic disorder, currently symptomatic major depressive disorder, schizophrenia
* History of exercise intolerance
* Any finding on examination indicative of cardiac or respiratory compromise
* History of heart disease
* History of pulmonary disease, other than controlled, non-exercise-induced asthma
* History of uncontrolled diabetes
* Resting heart rate > 100 BPM
* Resting systolic blood pressure > 140 mmHg or diastolic blood pressure > 100 mmHg
* Peripheral condition making completion of the exercise protocol impossible, such as severe osteoarthritis or chronic pain
* Pregnancy
* For healthy subjects undergoing MRI:

  * Ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, or ocular foreign body
  * Implanted cardiac pacemaker or auto-defibrillator or pump
  * Non-removable body piercing
  * Claustrophobia
  * Inability to lie supine for two hours
  * Any structural brain abnormality, such as tumor or stroke

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-08-31; Primary Completion 2015-05-21 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Recall of pictures | 2 years

SECONDARY OUTCOMES:
Recall of word lists | 2 years
Digit-symbol substitution performance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Wassermann, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahlskog JE, Geda YE, Graff-Radford NR, Petersen RC. Physical exercise as a preventive or disease-modifying treatment of dementia and brain aging. Mayo Clin Proc. 2011 Sep;86(9):876-84. doi: 10.4065/mcp.2011.0252. PMID 21878600
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831